CLINICAL TRIAL: NCT04540783
Title: The Effects of Transcranial Direct Current Stimulation (tDCS) and Cognitive Training on Episodic Memory and Attention in Patients With Traumatic Brain Injury: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: The Effects of Transcranial Direct Current Stimulation (tDCS) and Cognitive Training in Patients With TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, WELLINGSON SILVA PAIVA, Supervisor, Division of Neurosurgery, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2241648
Record Dates: First submitted 2020-03-09; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Traumatic Brain Injury; Closed Traumatic Brain Injury; Severe Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: sham device (by code)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - G1 (Active Comparator): bitemporal anodal stimulation and cathodal stimulation at supraorbital region.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Group 2 - G2 (Active Comparator): dorsolateral prefrontal anodal stimulation and cathodal stimulation at contralateral supraorbital region.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Group 3 - G3 (Sham Comparator): sham anodal stimulation over bitemporal or dorsolateral prefrontal cortex (randomized) and sham cathodal over the orbitofrontal region.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — 10 sessions of 2mA and 20 minutes tDCS. Sponges size 5x7 cm. For the sham condition, the patient will receive just 30 seconds of stimulation.

SUMMARY:
Long-term sequelae in TBI is a well-recognized burn. We designed a proof of concept study, randomized, double-blind, placebo-controlled to evaluate 36 adult TBI patients. To evaluate the early and late effects of 10 days of 20 minutes applying transcranial direct-current stimulation (tDCS) in the dorsolateral prefrontal cortex (DLPFC), bilateral temporal cortex (CTB) and compare to sham stimulation, and online cognitive training. We expect that the active group will differ from the sham group, showing larger effect sizes in the cognitive assessment.

DETAILED DESCRIPTION:
Method: proof of concept study, randomized, double-blind, placebo-controlled. 36 adult patients will be recruited, with closed TBI for at least 6 months, of both sexes. The sequence of randomization will provide the allocation 1: 1: 1 in parallel groups: G1 n = 12 active (CTB), G2 n = 12 active (DLPFC), and G3 n = 12 (Sham). The tDCS will be held with the intensity of 2 mA for 20 minutes per session and online cognitive training (concurrent with the ETCC). All patients, after the screening and randomization, will make a baseline neuropsychological assessment (T0) and receive 10 sessions of stimulation concomitant to cognitive training. Patients will undergo neuropsychological reassessment one week (T1) and two months (T2) after the last tDCS session. We will evaluate performance on episodic memory tests, working memory and attention in the three periods (T0, T1, and T2). The significance adopted is the level of 5% (α = 0.05), analysis of 80% power and bicaudal curve. Analysis of the results will be done by intention to treat (ITT).

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis closed traumatic brain injury, cognitive complaints reported by the patient or caregiver.

Exclusion Criteria:

metal implants in the head, seizures, abnormal EEG, depressive symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Episodic Memory measured by The Rey Auditory-Verbal Learning Test (RAVLT) | up to 2 weeks
  List of words

SECONDARY OUTCOMES:
Memory cognitive training | up to 2 weeks
  The patients will receive 10 days of episodic memory training.
Attention cognitive training | up to 2 weeks
  The patients will receive 10 days of attention training.

OTHER OUTCOMES:
electroencephalogram - EEG | up to 2 weeks
  electroencephalogram will be used for safety (Alpha and delta wave)

CONTACTS AND LOCATIONS:
Overall Officials: Welligson S Paiva, MD PhD, Principal Investigator — professor
Locations (1):
- Faculdade de Medicina do Hospital das Clinicas HC-FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We need to discuss between the researchers.

REFERENCES:
- [Derived] De Freitas DJ, De Carvalho D, Paglioni VM, Brunoni AR, Valiengo L, Thome-Souza MS, Guirado VMP, Zaninotto AL, Paiva WS. Effects of transcranial direct current stimulation (tDCS) and concurrent cognitive training on episodic memory in patients with traumatic brain injury: a double-blind, randomised, placebo-controlled study. BMJ Open. 2021 Aug 26;11(8):e045285. doi: 10.1136/bmjopen-2020-045285. PMID 34446480